CLINICAL TRIAL: NCT03215277
Title: A Multicenter, Phase 2A, Randomized, Investigator-Blind, Subject-Blind, Parallel-Group Study to Evaluate the Efficacy and Safety of Bimekizumab and Certolizumab Pegol in Subjects With Active Ankylosing Spondylitis
Brief Title: A Study to Test the Efficacy and Safety of Bimekizumab and Certolizumab Pegol in Patients With Active Ankylosing Spondylitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AS0013; 2017-000957-37 (EudraCT Number)
Expanded Access: NCT03559686 (Available)
Record Dates: First submitted 2017-07-05; First posted 2017-07-12 (Actual); Results first posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Ankylosing Spondylitis
Keywords: Ankylosing Spondylitis; Bimekizumab; AS; Certolizumab Pegol; Cimzia
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — bimekizumab; Certolizumab Pegol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is an investigator-blind and subject-blind study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bimekizumab (Experimental): Subjects will receive several bimekizumab administrations on pre-defined time points. Placebo will be provided in this arm to mask the certolizumab pegol loading dose.
  Interventions: Drug: Bimekizumab; Other: Placebo
- Certolizumab pegol (Experimental): Subjects will receive several certolizumab pegol administrations on pre-defined time points.
  Interventions: Drug: Certolizumab pegol

INTERVENTIONS:
Drug: Bimekizumab — One bimekizumab dose will be administered.
  Other Names: UCB4940; BKZ
  Arms: Bimekizumab
Drug: Certolizumab pegol — Two certolizumab pegol doses will be administered. One of these doses is a loading dose.
  Other Names: CZP; Cimzia; CDP870
  Arms: Certolizumab pegol
Other: Placebo — Placebo will be provided to maintain the blinding.
  Arms: Bimekizumab

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of bimekizumab compared to certolizumab pegol in the treatment of subjects with active ankylosing spondylitis (AS).

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of active adult-onset ankylosing spondylitis (AS) as defined by documented radiologic evidence (X-ray) fulfilling the Modified New York criteria for AS (1984) of at least 3 months' symptom duration and age of onset <45 years
* Subject has moderate to severe active disease at the Screening Visit as defined by each of the following:

  1. Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) score >=4
  2. Spinal pain >=4 on a 0 to 10 numeric rating scale (NRS) (from BASDAI Item 2)
* Subjects must have had an inadequate response to, have a contraindication to, or have been intolerant to at least 2 nonsteroidal anti-inflammatory drugs (NSAIDs)
* Subjects taking corticosteroids must be on a maximum daily dose of <=10mg/day oral prednisolone or equivalent
* Subjects taking methotrexate (MTX; <=25 mg/week) are allowed to continue their medication if they received a stable dose for at least 12 weeks before randomization
* Subjects taking sulfasalazine (up to 3 grams/day) or hydroxychloroquine (up to 400 mg per day total) are allowed to continue their medication if started at least 12 weeks prior to randomization
* Subject who has been on an anti-tumor necrosis factor alpha (TNFα) agent must have experienced an inadequate response to previous or current treatment given at an approved dose for at least 3 months or have been intolerant to at least 1 administration of an anti-TNFα agent. Subjects may not have been on more than 1 anti-TNFα agent
* Subject has high-sensitive C-Reactive Protein (hsCRP) levels >=3 mg/L at the Screening Visit
* Female subjects must be postmenopausal, permanently sterilized or, if of childbearing potential, must be willing to use a highly effective method of contraception up till 20 weeks after last administration of investigational medicinal product (IMP)
* Male subjects with a partner of childbearing potential must be willing to use a condom when sexually active, up till 20 weeks after the last administration of IMP

Exclusion Criteria:

* Subject has received previous or current biological treatment other than TNFα inhibitor treatment
* Subjects with a total ankylosis of the spine, or a diagnosis of any other inflammatory arthritis eg, rheumatoid arthritis (RA), sarcoidosis, systemic lupus erythematosus, or reactive arthritis
* Subjects with any current sign or symptom that may indicate an active infection (except for the common cold)
* Subject has received previous or current biological treatment other than TNFα inhibitor treatment
* Subject has chronic, recurrent, recent serious / life-threatening or current infection, as defined in the protocol
* Subject has history of certain atypical infections, viral hepatitides, human immunodeficiency virus (HIV) infection, tuberculosis, as defined in the protocol
* Subjects receiving any live vaccination within the 8 weeks prior to Baseline
* Subjects with known tuberculosis (TB) infection, at high risk of acquiring TB infection, with latent TB infection or current or history of nontuberculous mycobacteria (NTMB) infection
* Subject has immunosuppressive condition or treatment, recent history of malignancy (some exceptions) or demyelinating disease
* Subjects with concurrent malignancy or a history of malignancy during the past 5 years will be excluded, with following exceptions that may be included:

  1. <= 3 excised or ablated basal cell carcinomas of the skin
  2. One squamous cell carcinoma of the skin (stage T1 maximum) successfully excised, or ablated only (other treatments, ie, chemotherapy, do not apply), with no signs of recurrence or metastases for more than 2 years prior to Screening
  3. Actinic keratosis (-es)
  4. Squamous cell carcinoma-in-situ of the skin successfully excised, or ablated, more than 6 months prior to Screening
* Subject has history of psychiatric disorder, including suicidality (as defined in the protocol
* Subject has major abnormalities on laboratory testing, as defined in the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2017-10-04 (Actual); Primary Completion 2020-05-25 (Actual); Study Completion 2020-05-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — +1-844-599-2273 (UCB)
Locations (34):
- United States (4):
  - As0013 908, Ormond Beach, Florida
  - As0013 903, Lincoln, Nebraska
  - As0013 902, Oklahoma City, Oklahoma
  - As0013 906, Memphis, Tennessee
- Czechia (4):
  - As0013 202, Kladno
  - As0013 205, Ostrava
  - As0013 201, Prague
  - As0013 203, Prague
- Germany (5):
  - As0013 302, Berlin
  - As0013 306, Berlin
  - As0013 304, Erlangen
  - As0013 303, Hamburg
  - As0013 301, Herne
- Greece (5):
  - As0013 405, Athens
  - As0013 404, Heraklion
  - As0013 401, Pátrai
  - As0013 402, Thessaloniki
  - As0013 406, Thessaloniki
- As0013 501, Chisinau, Moldova
- As0013 601, Amsterdam, Netherlands
- Poland (8):
  - As0013 708, Bialystok
  - As0013 709, Krakow
  - As0013 706, Olsztyn
  - As0013 703, Poznan
  - As0013 702, Torun
  - As0013 701, Warsaw
  - As0013 704, Warsaw
  - As0013 707, Wroclaw
- Russia (6):
  - As0013 801, Kazan'
  - As0013 803, Kemerovo
  - As0013 806, Moscow
  - As0013 807, Moscow
  - As0013 802, Yaroslavl
  - As0013 805, Yaroslavl

IPD SHARING:
Plan to Share IPD: Yes
Data from this study may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.clinicalstudydatarequest.com and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal. This plan may change if a determination is made that the data cannot be adequately anonymized.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this study may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.clinicalstudydatarequest.com and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Baraliakos X, de Jongh J, Poddubnyy D, Zwezerijnen GJC, Hemke R, Glatt S, Shaw S, Ionescu L, El Baghdady A, Mann J, Maguire RP, Vaux T, de Peyrecave N, Oortgiesen M, Baeten D, van der Laken C. Impact of bimekizumab and certolizumab pegol on efficacy, safety and osteoblastic activity in radiographic axial spondyloarthritis: results from a phase IIa, multicentre, randomised, double-blind, exploratory study with PET-CT imaging. Ther Adv Musculoskelet Dis. 2024 Nov 28;16:1759720X241293944. doi: 10.1177/1759720X241293944. eCollection 2024. PMID 39620046
- See also: Product Information — https://www.ucb.com/_up/ucb_com_products/documents/Cimzia_01_03_2023_en.pdf
- See also: Product Information — https://www.ema.europa.eu/en/documents/product-information/bimzelx-epar-product-information_en.pdf
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll study participants in October 2017 and concluded in May 2020.
Pre-assignment Details: The Participant Flow refers to the Randomized Set (RS).
Groups:
- Certolizumab Pegol: Participants received certolizumab pegol (CZP) 400 milligrams (mg) subcutaneously (sc) every 2 weeks (Q2W) at Weeks 0, 2, and 4 (loading dose) followed by CZP 200 mg sc Q2W in Weeks 6 to 10 and 400 mg every 4 weeks (Q4W) from Week 12 to Week 44.
- Bimekizumab: Participants received bimekizumab (BKZ) 160 mg sc Q2W from Week 0 through Week 10 and 320 mg sc Q4W from Week 12 to Week 44. In addition, participants received placebo injection to maintain the blind for the CZP loading dose at Baseline, Week 2 and Week 4.
Period: Overall Study
Arm/Group | Certolizumab Pegol | Bimekizumab
Started | 25 | 51
Completed | 22 | 46
Not Completed | 3 | 5
Not completed — Adverse Event | 2 | 3
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Participant was unable to attend clinic visit | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to Safety Set which consisted of all randomized study participants who received at least 1 dose (full or partial) of the investigational medicinal product (IMP).
Arm/Group | Certolizumab Pegol | Bimekizumab | Total Title
Number analyzed (Participants) | 25 | 51 | 76
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 47 | 72
  >=65 years | 0 | 4 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.7 (8.2) | 40.3 (12.5) | 40.1 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 11
  Male | 21 | 44 | 65
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 25 | 51 | 76
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 25 | 51 | 76

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Ankylosing Spondylitis Disease Activity Score (ASDAS) at Week 12
Description: ASDAS was calculated as the sum of the results from the following components: 0.121xTotal spinal pain (Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) Question 2 result), 0.058xDuration of morning stiffness (BASDAI Question 6 result), 0.110xPGADA, 0.073xPeripheral pain/swelling (BASDAI Question 3 result), 0.579x(natural logarithm of the CRP [mg/L] + 1), Spinal pain, PGADA, duration of morning stiffness, peripheral pain/swelling were all assessed on a numerical scale (0 to 10 units). There is a minimum score of 0.980 for ASDAS (as a fixed value of 2 was assumed for values of hs-CRP below the LLOQ), but no defined upper score. The change from Baseline is calculated, a negative value indicating improvement and a positive value worsening. Posterior means and 95% credible intervals in each group are presented.
Time Frame: From Baseline to Week 12
Population: Per Protocol Set (PPS) consisted of all study participants in the Full Analysis Set who had no important protocol deviation affecting the primary efficacy variable. Here, Number of participants analyzed signifies those participants who were evaluable for this outcome measure.
Measure: Mean (95% Confidence Interval); unit: scores on a scale
Groups:
- Certolizumab Pegol (PPS): Participants received CZP 400 mg sc Q2W at Weeks 0, 2, and 4 (loading dose) followed by CZP 200 mg sc Q2W in Weeks 6 to 10 and 400 mg Q4W from Week 12 to Week 44. Participants formed the Per Protocol Set (PPS).
- Bimekizumab (PPS): Participants received BKZ 160 mg sc Q2W from Week 0 through Week 10 and 320 mg sc Q4W from Week 12 to Week 44. In addition, participants received placebo injection to maintain the blind for the CZP loading dose at Baseline, Week 2 and Week 4. Participants formed the PPS.
Arm/Group | Certolizumab Pegol (PPS) | Bimekizumab (PPS)
Number analyzed (Participants) | 24 | 46
scores on a scale | -1.83 [-2.11 to -1.55] | -2.06 [-2.30 to -1.81]
Statistical Analysis 1: Comparison: Certolizumab Pegol (PPS) vs Bimekizumab (PPS); Results were based on a complete case (ie, data as observed) Bayesian linear model with the change from Baseline in ASDAS as the independent variable. Treatment was included as a predictor in the model and Baseline ASDAS as a covariate. The mean posterior difference and 95% credible interval were presented for the BKZ vs CZP comparison; Test type: Superiority; Regression, Linear; Mean Posterior Difference = 0.23, 95% CI 2-sided [-0.14 to 0.60]
Statistical Analysis 2: Comparison: Certolizumab Pegol (PPS) vs Bimekizumab (PPS); Results were based on a complete case (ie, data as observed) Bayesian linear model with the change from Baseline in ASDAS as the independent variable. Treatment was included as a predictor in the model and Baseline ASDAS as a covariate. Pr[Diff>0%](%) refers to the probability that the mean change from Baseline in ASDAS in the BKZ group was greater than the mean change from Baseline in ASDAS in the CZP group; Test type: Superiority; Regression, Linear; PR[Diff > 0%](%) = 88.4

2. Primary Outcome: Number of Participants With Adverse Events (AE) During the Study Conduct
Description: An AE was any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. A treatment-emergent adverse event (TEAE) was defined as any AE with a start date/time at the time of or after the first dose of IMP up until 140 days after the last dose of IMP.
Time Frame: From Baseline until Safety Follow-Up Visit (up to Week 64)
Population: Safety Set (SS) consisted of all randomized study participants who received at least 1 dose (full or partial) of the IMP.
Measure: Count of Participants; unit: Participants
Groups:
- Certolizumab Pegol (SS): Participants received CZP 400 mg sc Q2W at Weeks 0, 2, and 4 (loading dose) followed by CZP 200 mg sc Q2W in Weeks 6 to 10 and 400 mg Q4W from Week 12 to Week 44. Participants formed the Safety Set (SS).
- Bimekizumab (SS): Participants received BKZ 160 mg sc Q2W from Week 0 through Week 10 and 320 mg sc Q4W from Week 12 to Week 44. In addition, participants received placebo injection to maintain the blind for the CZP loading dose at Baseline, Week 2 and Week 4. Participants formed the SS.
Arm/Group | Certolizumab Pegol (SS) | Bimekizumab (SS)
Number analyzed (Participants) | 25 | 51
Participants | 19 | 42

3. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs) During the Study Conduct
Description: An SAE was any untoward medical occurrence that at any dose: - Resulted in death - Is life-threatening - Required in patient hospitalisation or prolongation of existing hospitalisation - Is a congenital anomaly or birth defect - Is an infection that requires treatment with parenteral antibiotics - Other important medical events which based on medical or scientific judgement may jeopardised the participants, or may require medical or surgical intervention to prevent any of the above. A TEAE was defined as any AE with a start date/time at the time of or after the first dose of IMP up until 140 days after the last dose of IMP.
Time Frame: From Baseline until Safety Follow-Up Visit (up to Week 64)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Certolizumab Pegol (SS) | Bimekizumab (SS)
Number analyzed (Participants) | 25 | 51
Participants | 3 | 5

4. Primary Outcome: Number of Participants Who Withdrew Due to an Adverse Event (AE) During the Study Conduct
Description: An AE was any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. A TEAE was defined as any AE with a start date/time at the time of or after the first dose of IMP up until 140 days after the last dose of IMP.
Time Frame: From Baseline until Safety Follow-Up Visit (up to Week 64)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Certolizumab Pegol (SS) | Bimekizumab (SS)
Number analyzed (Participants) | 25 | 51
Participants | 3 | 3

5. Secondary Outcome: Number of Participants With Ankylosing Spondylitis Disease Activity Score - Inactive Disease (ASDAS-ID) at Week 12
Description: ASDAS-ID was defined by ASDAS < 1.3. ASDAS was calculated as the sum of the results from the following components: 0.121xTotal spinal pain (Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) Question 2 result), 0.058xDuration of morning stiffness (BASDAI Question 6 result), 0.110xPGADA, 0.073xPeripheral pain/swelling (BASDAI Question 3 result), 0.579x(natural logarithm of the CRP [mg/L] + 1), Spinal pain, PGADA, duration of morning stiffness, peripheral pain/swelling were all assessed on a numerical scale (0 to 10 units). There is a minimum score of 0.980 for ASDAS (as a fixed value of 2 was assumed for values of hs-CRP below the LLOQ), but no defined upper score.
Time Frame: Week 12
Population: Per-Protocol Set (PPS) consisted of all study participants in the Full Analysis Set who had no important protocol deviation affecting the primary efficacy variable. Here, Number of participants analyzed signifies those participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Certolizumab Pegol (PPS) | Bimekizumab (PPS)
Number analyzed (Participants) | 24 | 46
Participants | 5 | 11

6. Secondary Outcome: Number of Participants With Ankylosing Spondylitis Disease Activity Score-Major Improvement (ASDAS-MI) at Week 12
Description: ASDAS-MI was defined by a reduction (improvement) from Baseline in ASDAS >=2 units. ASDAS was calculated as the sum of the results from the following components: 0.121xTotal spinal pain (Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) Question 2 result), 0.058xDuration of morning stiffness (BASDAI Question 6 result), 0.110xPGADA, 0.073xPeripheral pain/swelling (BASDAI Question 3 result), 0.579x(natural logarithm of the CRP [mg/L] + 1), Spinal pain, PGADA, duration of morning stiffness, peripheral pain/swelling were all assessed on a numerical scale (0 to 10 units). There is a minimum score of 0.980 for ASDAS (as a fixed value of 2 was assumed for values of hs-CRP below the LLOQ), but no defined upper score.
Time Frame: Baseline, Week 12
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Certolizumab Pegol (PPS) | Bimekizumab (PPS)
Number analyzed (Participants) | 24 | 46
Participants | 11 [27.9 to 64.9] | 28 [46.5 to 73.6]

ADVERSE EVENTS:
Time Frame: From Baseline until Safety Follow-Up Visit (up to Week 64)
Description: A treatment-emergent adverse event (TEAE) was defined as any AE with a start date/time at the time of or after the first dose of IMP up until 140 days after the last dose of IMP.
Arm/Group | Certolizumab Pegol (SS) | Bimekizumab (SS)
All-Cause Mortality (participants affected / at risk) | 1/25 | 0/51
Serious Adverse Events (participants affected / at risk) | 3/25 | 5/51
Other Adverse Events (participants affected / at risk) | 16/25 | 27/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Certolizumab Pegol (SS) (N=25) | Bimekizumab (SS) (N=51)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Uveitis (Eye disorders) | 0 (0) | 1 (1)
Arthritis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (2)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Traumatic arthritis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Myasthenia gravis (Nervous system disorders) | 1 (1) | 0 (0)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Certolizumab Pegol (SS) (N=25) | Bimekizumab (SS) (N=51)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 6 (8)
Oral herpes (Infections and infestations) | 2 (2) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 3 (4)
Nasopharyngitis (Infections and infestations) | 6 (8) | 10 (12)
Pharyngitis (Infections and infestations) | 0 (0) | 5 (5)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 3 (3)
Tonsillitis (Infections and infestations) | 2 (2) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 3 (5)
Alanine aminotransferase increased (Investigations) | 2 (3) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 2 (5) | 1 (2)
Periarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4)
Headache (Nervous system disorders) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-02-27): https://cdn.clinicaltrials.gov/large-docs/77/NCT03215277/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-19): https://cdn.clinicaltrials.gov/large-docs/77/NCT03215277/SAP_001.pdf